CLINICAL TRIAL: NCT00174915
Title: A Phase 3, Randomized, Multicenter, Allopurinol and Placebo-Controlled Study Assessing the Safety and Efficacy of Oral Febuxostat in Subjects With Gout.
Brief Title: Phase 3, Febuxostat, Allopurinol and Placebo-Controlled Study in Gout Subjects.
Acronym: APEX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C02-009; U1111-1113-9740 (Registry Identifier: WHO)
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Results first posted 2009-07-16 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Gout
Keywords: Uric Acid, gout, xanthine oxidase, febuxostat, tophi
MeSH Terms: conditions — Gout | interventions — Febuxostat; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Febuxostat 80 mg QD (Experimental)
  Interventions: Drug: Febuxostat
- Febuxostat 120 mg QD (Experimental)
  Interventions: Drug: Febuxostat
- Febuxostat 240 mg QD (Experimental)
  Interventions: Drug: Febuxostat
- Allopurinol QD (Active Comparator)
  Interventions: Drug: Allopurinol
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Febuxostat — Febuxostat 80 mg, orally, once daily for up to 28 weeks.
  Other Names: TMX-67; Tei-6720; Uloric
  Arms: Febuxostat 80 mg QD
Drug: Febuxostat — Febuxostat 120 mg, orally, once daily for up to 28 weeks.
  Other Names: TMX-67; Tei-6720; Uloric
  Arms: Febuxostat 120 mg QD
Drug: Febuxostat — Febuxostat 240 mg, orally, once daily for up to 28 weeks.
  Other Names: TMX-67; Tei-6720; Uloric
  Arms: Febuxostat 240 mg QD
Drug: Allopurinol — Allopurinol, orally, once daily for up to 28 weeks. Dose of allopurinol received was based on renal status. Subjects with serum creatinine ≤1.5 mg/dL received 300 mg once daily; subjects with serum creatinine >1.5 mg/dL and ≤2.0 mg/dL received 100 mg once daily.
  Arms: Allopurinol QD
Drug: Placebo — Placebo, orally, once daily for up to 28 weeks.
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to compare febuxostat, allopurinol and placebo, once daily (QD), in subjects with gout.

DETAILED DESCRIPTION:
A Phase 3 Study comparing 80 mg, 120 mg or 240 mg of febuxostat, allopurinol (300 mg for those with normal renal function and 100 mg for those with impaired renal function) and placebo administered once daily in subjects with gout.

Subjects will receive treatment for 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Hyperuricemia (serum urate ≥8.0 mg/dL and gout by American Rheumatism Association Criteria
* Renal function defined as a serum creatinine level of < 2.0 mg/dL and creatinine clearance of > 20 milliliters per minute (mL/min) by Cockroft and Gault formula.

Exclusion Criteria:

* History of xanthinuria
* Intolerance to allopurinol
* Presence of renal calculi,
* Alcohol intake of ≥ 14 drinks/week
* Clinically significant medical condition

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1072 (Actual)
Dates: Start 2003-02; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda

REFERENCES:
- [Result] Schumacher HR Jr, Becker MA, Wortmann RL, Macdonald PA, Hunt B, Streit J, Lademacher C, Joseph-Ridge N. Effects of febuxostat versus allopurinol and placebo in reducing serum urate in subjects with hyperuricemia and gout: a 28-week, phase III, randomized, double-blind, parallel-group trial. Arthritis Rheum. 2008 Nov 15;59(11):1540-8. doi: 10.1002/art.24209. PMID 18975369
- [Result] Becker MA, MacDonald PA, Hunt BJ, Lademacher C, Joseph-Ridge N. Determinants of the clinical outcomes of gout during the first year of urate-lowering therapy. Nucleosides Nucleotides Nucleic Acids. 2008 Jun;27(6):585-91. doi: 10.1080/15257770802136032. PMID 18600509
- [Result] Wortmann RL, Macdonald PA, Hunt B, Jackson RL. Effect of prophylaxis on gout flares after the initiation of urate-lowering therapy: analysis of data from three phase III trials. Clin Ther. 2010 Dec;32(14):2386-97. doi: 10.1016/j.clinthera.2011.01.008. PMID 21353107
- [Result] Chohan S, Becker MA, MacDonald PA, Chefo S, Jackson RL. Women with gout: efficacy and safety of urate-lowering with febuxostat and allopurinol. Arthritis Care Res (Hoboken). 2012 Feb;64(2):256-61. doi: 10.1002/acr.20680. PMID 22052584
- See also: Uloric Package Insert — http://general.takedapharm.com/content/file.aspx?applicationcode=6C7C39D8-5D09-453B-BF30-696A4AB88E62&fileTypeCode=ULORICPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 167 investigative sites in the United States from 21 February 2003 to 07 April 2004.
Pre-assignment Details: Subjects currently receiving urate-lowering therapy discontinued those urate-lowering therapies and initiated prophylactic medications before enrollment in once daily (QD) treatment groups.
Groups:
- Febuxostat 80 mg QD: Febuxostat 80 mg, orally, once daily for up to 28 weeks.
- Febuxostat 120 mg QD: Febuxostat 120 mg, orally, once daily for up to 28 weeks.
- Febuxostat 240 mg QD: Febuxostat 240 mg, orally, once daily for up to 28 weeks.
- Allopurinol QD: Allopurinol, orally, once daily for up to 28 weeks. Dose of allopurinol received was based on renal status. Subjects with serum creatinine ≤1.5 mg/dL received 300 mg once daily; subjects with serum creatinine >1.5 mg/dL and ≤2.0 mg/dL received 100 mg once daily.
- Placebo QD: Placebo, orally, once daily for up to 28 weeks.
Period: Overall Study
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Febuxostat 240 mg QD | Allopurinol QD | Placebo QD
Started | 267 | 269 | 134 | 268 | 134
Completed | 174 | 200 | 86 | 211 | 101
Not Completed | 93 | 69 | 48 | 57 | 33
Not completed — Lost to Follow-up | 19 | 17 | 9 | 17 | 10
Not completed — Adverse Event | 18 | 16 | 11 | 18 | 5
Not completed — Personal Reason(s) | 16 | 16 | 9 | 9 | 9
Not completed — Other | 15 | 8 | 6 | 5 | 3
Not completed — Gout Flare | 13 | 6 | 8 | 1 | 0
Not completed — Protocol Violation | 6 | 3 | 3 | 6 | 3
Not completed — Therapeutic Failure | 6 | 3 | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Febuxostat 240 mg QD | Allopurinol QD | Placebo QD | Total
Number analyzed (Participants) | 267 | 269 | 134 | 268 | 134 | 1072
Age, Customized [Number; unit: subjects]
  <45 years | 82 | 79 | 33 | 82 | 36 | 312
  45 years to <65 years | 146 | 154 | 71 | 147 | 79 | 597
  ≥65 years | 39 | 36 | 30 | 39 | 19 | 163
Age Continuous [Mean (Standard Deviation); unit: years] | 50.6 (12.24) | 51.2 (11.57) | 54.3 (12.83) | 51.8 (12.25) | 51.5 (12.18) | 51.6 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 8 | 19 | 11 | 67
  Male | 251 | 256 | 126 | 249 | 123 | 1005
Race/Ethnicity, Customized [Number; unit: subjects]
  White | 200 | 214 | 107 | 206 | 108 | 835
  Black or African American | 38 | 27 | 13 | 33 | 9 | 120
  Hispanic | 13 | 16 | 8 | 17 | 10 | 64
  Asian | 8 | 8 | 1 | 6 | 3 | 26
  Other | 8 | 4 | 5 | 6 | 4 | 27
Body Mass Index [Number; unit: subjects]
  <18.5 kilogram per meter² (kg/m²) | 0 | 0 | 0 | 0 | 0 | 0
  18.5 kg/m² to <25 kg/m² | 10 | 11 | 9 | 15 | 16 | 61
  25 kg/m² to <30 kg/m² | 85 | 81 | 42 | 91 | 48 | 347
  ≥30 kg/m² | 172 | 176 | 83 | 161 | 70 | 662
  missing | 0 | 1 | 0 | 1 | 0 | 2
Presence of a Primary PalpableTophus [Number; unit: subjects]
  Yes | 48 | 53 | 25 | 64 | 29 | 219
  No, but other tophi present | 0 | 3 | 1 | 1 | 1 | 6
  No, and no other tophi present | 219 | 213 | 108 | 203 | 104 | 847
Serum Creatinine [Number; unit: subjects]
  ≤1.5 milligram per deciliter (mg/dL) | 258 | 258 | 129 | 258 | 129 | 1032
  >1.5 mg/dL | 9 | 11 | 5 | 10 | 5 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Whose Last Three Serum Urate Levels Are <6.0 Milligram Per Deciliter (mg/dL).
Description: Each subject's serum urate at the last 3 visits determined the subject's response for the primary efficacy variable. A subject who prematurely discontinued without least 3 postbaseline serum urate levels was considered a nonresponder; if at least 3 serum urate were obtained postbaseline, those 3 visits were used. The last 3 visits used may have differed for each subject.
Time Frame: Last 3 visits (any last 3 visits up to week 28)
Population: Analysis was performed on all randomized subjects who took at least 1 dose of study drug and had a baseline serum urate ≥8.0 mg/dL. If subject prematurely discontinued from study before at least 3 serum urate levels were obtained, subject was considered a nonresponder; if at least 3 serum urate were obtained postbaseline, those 3 visits were used.
Measure: Number; unit: Percentage of subjects
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Febuxostat 240 mg QD | Allopurinol QD | Placebo QD
Number analyzed (Participants) | 262 | 269 | 134 | 268 | 134
Percentage of subjects | 48 | 65 | 69 | 22 | 0
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The overall 0.05 level of significance for the multiple comparisons of each febuxostat dose to placebo was controlled using Hochberg's method. The p-value was statistically significant; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL versus [v.] >1.5 mg/dL)
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 3: Comparison: Febuxostat 240 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 4: Comparison: Febuxostat 80 mg QD vs Allopurinol QD; Test type: Non-Inferiority or Equivalence — Non-inferiority of febuxostat 80 mg to allopurinol was declared if the value of the lower bound of the 97.5% confidence interval is > -10%; Difference in percentage = 25.7, 97.5% CI [16.7 to 34.7]
Statistical Analysis 5: Comparison: Febuxostat 120 mg QD vs Allopurinol QD; Test type: Non-Inferiority or Equivalence — Non-inferiority of febuxostat 120 mg to allopurinol was declared if the value of the lower bound of the 97.5% confidence interval is > -10%; Difference in percentage = 42.7, 97.5% CI [34.0 to 51.3]
Statistical Analysis 6: Comparison: Febuxostat 80 mg QD vs Allopurinol QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Comparisons of each febuxostat dose to allopurinol were adjusted to control the overall 0.05 level of significance for superiority by using Hochberg's method. The p-value was statistically significant; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 7: Comparison: Febuxostat 120 mg QD vs Allopurinol QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 6]; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 8: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 9: Comparison: Febuxostat 240 mg QD vs Allopurinol QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 10: Comparison: Febuxostat 80 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 11: Comparison: Febuxostat 120 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p = 0.479, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 12: Comparison: Allopurinol QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)

2. Secondary Outcome: Percentage of Subjects Whose Serum Urate Levels Are <6.0 mg/dL at Week 28
Description: Serum urate values were obtained at the Week 28 visit. The percentage of subjects whose serum urate was <6.0 mg/dL at the Week 28 visit was summarized.
Time Frame: Week 28
Population: Analysis was performed on intend to treat (ITT) subjects, which were defined as all randomized subjects who took at least 1 dose of study drug and who had a baseline serum urate ≥8.0 mg/dL. Missing data were not imputed.
Measure: Number; unit: Percentage of subjects
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Febuxostat 240 mg QD | Allopurinol QD | Placebo QD
Number analyzed (Participants) | 161 | 188 | 83 | 208 | 99
Percentage of subjects | 76 | 87 | 94 | 41 | 1
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 3: Comparison: Febuxostat 240 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 4: Comparison: Febuxostat 80 mg QD vs Allopurinol QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 5: Comparison: Febuxostat 120 mg QD vs Allopurinol QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 6: Comparison: Febuxostat 240 mg QD vs Allopurinol QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 7: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p = 0.011, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 8: Comparison: Febuxostat 80 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 9: Comparison: Febuxostat 120 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p = 0.091, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 10: Comparison: Allopurinol QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)

3. Secondary Outcome: Percentage of Subjects Whose Serum Urate Levels Are <6.0 mg/dL at Final Visit
Description: The percentage of subjects whose serum urate was <6.0 mg/dL at the final visit was summarized. The final visit was the last visit at which a serum urate value was collected and may have differed by subject.
Time Frame: Final Visit (up to 28 weeks).
Population: Analysis was performed on the ITT subjects, which were defined as all randomized subjects who took at least 1 dose of study drug and who had a baseline serum urate ≥8.0 mg/dL. Missing data were not imputed.
Measure: Number; unit: Percentage of subjects
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Febuxostat 240 mg QD | Allopurinol QD | Placebo QD
Number analyzed (Participants) | 253 | 265 | 126 | 263 | 127
Percentage of subjects | 72 | 79 | 92 | 39 | 1
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 3: Comparison: Febuxostat 240 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 4: Comparison: Febuxostat 80 mg QD vs Allopurinol QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 5: Comparison: Febuxostat 120 mg QD vs Allopurinol QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 6: Comparison: Febuxostat 240 mg QD vs Allopurinol QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 7: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p = 0.074, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 8: Comparison: Febuxostat 80 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 9: Comparison: Febuxostat 120 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 10: Comparison: Allopurinol QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)

4. Secondary Outcome: Percent Change From Baseline in Serum Urate Levels at Week 28.
Description: Serum urate values were obtained at the Week 28 visit. The percent change in serum urate was calculated as [(Week 28 - baseline levels)/baseline]*100 and summarized.
Time Frame: Baseline and Week 28
Population: Analysis was performed on the ITT subjects, which were defined as all randomized subjects. who took at least 1 dose of study drug and who had a baseline serum urate ≥8.0 mg/dL. Missing data were not imputed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Febuxostat 240 mg QD | Allopurinol QD | Placebo QD
Number analyzed (Participants) | 161 | 188 | 83 | 208 | 99
Percent change | -47.6 (15.86) | -54.9 (14.97) | -67.8 (18.18) | -34.4 (14.21) | -3.6 (13.85)
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANOVA — P-values for pairwise comparisons are from contrast within the framework of the ANOVA model with treatment and baseline renal function as factors. Statistical significance was determined at the 0.05 level without adjustments for multiple comparisons
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 240 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Febuxostat 80 mg QD vs Allopurinol QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Febuxostat 120 mg QD vs Allopurinol QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Febuxostat 240 mg QD vs Allopurinol QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: Febuxostat 80 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 9: Comparison: Febuxostat 120 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 10: Comparison: Allopurinol QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]

5. Secondary Outcome: Percent Change From Baseline in Serum Urate Levels at Final Visit
Description: The percent change in serum urate from baseline to the Final visit was summarized. The percent change in serum urate was calculated as [(Final visit - baseline levels)/baseline]*100. The final visit was the last visit at which a serum urate value was collected. The timing of the final visit may have differed for each subject.
Time Frame: Baseline and Final Visit (up to 28 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Febuxostat 240 mg QD | Allopurinol QD | Placebo QD
Number analyzed (Participants) | 253 | 265 | 126 | 263 | 127
Percent change | -45.2 (18.16) | -51.9 (17.99) | -66.3 (20.62) | -33.7 (14.75) | -3.0 (13.28)
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 240 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Febuxostat 80 mg QD vs Allopurinol QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Febuxostat 120 mg QD vs Allopurinol QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Febuxostat 240 mg QD vs Allopurinol QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: Febuxostat 80 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 9: Comparison: Febuxostat 120 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 10: Comparison: Allopurinol QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 4, analysis 1]

6. Secondary Outcome: Percent Change in Primary Tophus Size at Week 28, as Determined by Physical Measurement in the Subset of Subjects With Palpable Tophi at the Screening Visit.
Description: The percent change from baseline in primary tophus size as determined by physical measurement was calculated as [(Week 28 - baseline sizes)/baseline]*100 for the subset of subjects with a primary palpable tophus at the Screening Visit. If the primary tophus was no longer palpable at the Week 28 visit, the size was assumed to be zero.
Time Frame: Baseline and Week 28
Population: Analysis was performed on the ITT subjects, which were defined as all randomized subjects who took at least 1 dose of study drug, who had a baseline serum urate ≥8.0 mg/dL, and who had a palpable primary tophus measured at baseline. Missing data were not imputed.
Measure: Median (Inter-Quartile Range); unit: percent change from baseline
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Febuxostat 240 mg QD | Allopurinol QD | Placebo QD
Number analyzed (Participants) | 26 | 35 | 14 | 46 | 21
percent change from baseline | -45.6 [-85.9 to 3.0] | -54.2 [-100.0 to -16.7] | -53.2 [-77.8 to -22.1] | -31.5 [-95.0 to 5.6] | -52.0 [-62.5 to -21.4]
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.789, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.320, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Febuxostat 240 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.381, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 4: Comparison: Febuxostat 80 mg QD vs Allopurinol QD; Test type: Superiority or Other; p = 0.809, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 5: Comparison: Febuxostat 120 mg QD vs Allopurinol QD; Test type: Superiority or Other; p = 0.154, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 6: Comparison: Febuxostat 240 mg QD vs Allopurinol QD; Test type: Superiority or Other; p = 0.247, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 7: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p = 0.415, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 8: Comparison: Febuxostat 80 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p = 0.649, Wilcoxon (Mann-Whitney) — Statistical significance was determined at the 0.05 level without adjustment for multiple comparisons
Statistical Analysis 9: Comparison: Febuxostat 120 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p = 0.807, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 10: Comparison: Allopurinol QD vs Placebo QD; Test type: Superiority or Other; p = 0.844, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons

7. Secondary Outcome: Percent Change in Primary Tophus Size at Final Visit, as Determined by Physical Measurement in the Subset of Subjects With Palpable Tophi at the Screening Visit.
Description: Percent change in primary tophus size was calculated as [(Final Visit - baseline sizes)/baseline]*100 for the subset of subjects with a primary palpable tophus at Screening. If tophus was not palpable at Final visit, the size was assumed to be 0. The timing of the final visit may have differed for each subject.
Time Frame: Baseline and Final Visit (up to 28 weeks)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: percent change from baseline
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Febuxostat 240 mg QD | Allopurinol QD | Placebo QD
Number analyzed (Participants) | 42 | 50 | 24 | 61 | 26
percent change from baseline | -33.8 [-85.4 to 0.0] | -42.4 [-90.3 to 0.0] | -47.0 [-80.0 to -13.8] | -22.6 [-66.7 to 0] | -40.3 [-62.5 to -16.7]
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.699, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.822, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Febuxostat 240 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.579, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 4: Comparison: Febuxostat 80 mg QD vs Allopurinol QD; Test type: Superiority or Other; p = 0.679, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 5: Comparison: Febuxostat 120 mg QD vs Allopurinol QD; Test type: Superiority or Other; p = 0.278, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 6: Comparison: Febuxostat 240 mg QD vs Allopurinol QD; Test type: Superiority or Other; p = 0.104, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 7: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p = 0.560, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 8: Comparison: Febuxostat 80 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p = 0.309, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 9: Comparison: Febuxostat 120 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p = 0.759, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 10: Comparison: Allopurinol QD vs Placebo QD; Test type: Superiority or Other; p = 0.385, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons

8. Secondary Outcome: Change in the Total Number of Tophi at Week 28 in the Subset of Subjects With Palpable Tophi at the Screening Visit.
Description: Change from baseline at Week 28 in the total number of tophi per subject was calculated for the subset of subjects with palpable tophi at the Screening Visit. If the tophi were not palpable at the Week 28 visit, the total count was assumed to be 0.
Time Frame: Baseline and Week 28
Population: Analysis was performed on the ITT subjects, which were defined as all randomized subjects who took at least 1 dose of study drug,had a baseline serum urate ≥8.0 mg/dL, and had palpable tophi at the screening visit. Missing data were not imputed.
Measure: Median (Inter-Quartile Range); unit: number of tophi
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Febuxostat 240 mg QD | Allopurinol QD | Placebo QD
Number analyzed (Participants) | 28 | 38 | 16 | 47 | 22
number of tophi | 0.0 [-0.5 to 0.0] | 0.0 [-2.0 to 0.0] | 0.0 [-1.0 to 0.0] | 0.0 [-1.0 to 0.0] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.949, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.050, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Febuxostat 240 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.577, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 4: Comparison: Febuxostat 80 mg QD vs Allopurinol QD; Test type: Superiority or Other; p = 0.598, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 5: Comparison: Febuxostat 120 mg QD vs Allopurinol QD; Test type: Superiority or Other; p = 0.062, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 6: Comparison: Febuxostat 240 mg QD vs Allopurinol QD; Test type: Superiority or Other; p = 0.969, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 7: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p = 0.056, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 8: Comparison: Febuxostat 80 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p = 0.659, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 9: Comparison: Febuxostat 120 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p = 0.197, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 10: Comparison: Allopurinol QD vs Placebo QD; Test type: Superiority or Other; p = 0.521, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons

9. Secondary Outcome: Change in the Total Number of Tophi at Final Visit in the Subset of Subjects With Palpable Tophi at the Screening Visit
Description: Change in number of tophi/subject was calculated for the subset of subjects with palpable tophi at the Screening. If the tophi were not palpable at the Final Visit, total count was assumed to be 0. The timing of the final visit may have differed for each subject.
Time Frame: Final Visit (up to 28 weeks)
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: number of tophi
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Febuxostat 240 mg QD | Allopurinol QD | Placebo QD
Number analyzed (Participants) | 42 | 53 | 25 | 62 | 27
number of tophi | 0.0 [0.0 to 0.0] | 0.0 [-1.0 to 0.0] | 0.0 [-1.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.683, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.078, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 3: Comparison: Febuxostat 240 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.442, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 4: Comparison: Febuxostat 80 mg QD vs Allopurinol QD; Test type: Superiority or Other; p = 0.990, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 5: Comparison: Febuxostat 120 mg QD vs Allopurinol QD; Test type: Superiority or Other; p = 0.077, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 6: Comparison: Febuxostat 240 mg QD vs Allopurinol QD; Test type: Superiority or Other; p = 0.662, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 7: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p = 0.139, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 8: Comparison: Febuxostat 80 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p = 0.705, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 9: Comparison: Febuxostat 120 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p = 0.337, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons
Statistical Analysis 10: Comparison: Allopurinol QD vs Placebo QD; Test type: Superiority or Other; p = 0.643, Wilcoxon (Mann-Whitney) — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons

10. Secondary Outcome: Percentage of Subjects Requiring Treatment for a Gout Flare Between Weeks 8 and 28 of the Double-Blind Treatment Period.
Description: Percentage of subjects requiring treatment for a gout flare between Weeks 8 and 28 of the double-blind treatment period was summarized. A subject who reported more than 1 gout flare during this period was counted only once.
Time Frame: Weeks 8 through 28
Population: Analysis was performed on the ITT subjects who had at least one dose of study drug between Weeks 8 and 28.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Febuxostat 240 mg QD | Allopurinol QD | Placebo QD
Number analyzed (Participants) | 223 | 240 | 106 | 237 | 119
percentage of subjects | 55 | 54 | 57 | 46 | 52
Statistical Analysis 1: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.645, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 2: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.756, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 3: Comparison: Febuxostat 240 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.428, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 4: Comparison: Febuxostat 80 mg QD vs Allopurinol QD; Test type: Superiority or Other; p = 0.076, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 5: Comparison: Febuxostat 120 mg QD vs Allopurinol QD; Test type: Superiority or Other; p = 0.106, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 6: Comparison: Febuxostat 240 mg QD vs Allopurinol QD; Test type: Superiority or Other; p = 0.069, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 7: Comparison: Febuxostat 80 mg QD vs Febuxostat 120 mg QD; Test type: Superiority or Other; p = 0.837, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 8: Comparison: Febuxostat 80 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p = 0.749, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 9: Comparison: Febuxostat 120 mg QD vs Febuxostat 240 mg QD; Test type: Superiority or Other; p = 0.581, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)
Statistical Analysis 10: Comparison: Allopurinol QD vs Placebo QD; Test type: Superiority or Other; p = 0.311, Cochran-Mantel-Haenszel — Statistical significance was determined at 0.05 level without adjustment for multiple comparisons; The Cochran-Mantel-Haenszel test was stratified by baseline renal function (serum creatinine ≤1.5 mg/dL v. >1.5 mg/dL)

ADVERSE EVENTS:
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Febuxostat 240 mg QD | Allopurinol QD | Placebo QD
Serious Adverse Events (participants affected / at risk) | 11/267 | 9/269 | 5/134 | 7/268 | 2/134
Other Adverse Events (participants affected / at risk) | 122/267 | 123/269 | 72/134 | 133/268 | 61/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Febuxostat 80 mg QD (N=267) | Febuxostat 120 mg QD (N=269) | Febuxostat 240 mg QD (N=134) | Allopurinol QD (N=268) | Placebo QD (N=134)
Anaemias not elsewhere classified (NEC) (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Cardiomyopathies (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary Artery Disorders NEC (Cardiac disorders) | 2 | 0 | 0 | 0 | 1
Ischaemic Coronary Artery Disorders (Cardiac disorders) | 1 | 2 | 0 | 0 | 0
Supraventricular Arrhythmias (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Abdominal Hernias, Site Unspecified (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Duodenal and Small Intestinal Stenosis and Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal & Abdominal Pain, Excluding Oral,Throat (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Intestinal Ulcers and Perforation NEC (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea and Vomiting Symptoms (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pain and Discomfort NEC (General disorders) | 2 | 1 | 0 | 1 | 0
Cholecystitis and Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Abdominal and Gastrointestinal Infections (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Device Failure and Malfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Device Related Complications (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Non-Site Specific Procedural Complications (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Hypoglycaemic Conditions NEC (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Total Fluid Volume Decreased (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Muscle Weakness Conditions (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteoarthropathies (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Colonic Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Endocrine Neoplasms Benign NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Endocrine Neoplasms Malignant and Unspecified NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Hodgkin's Disease NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Prostatic Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Seizures and Seizure Disorders NEC (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Transient Cerebrovascular Events (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Renal Failure and Impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Bronchospasm and Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Lower Respiratory Tract Signs and Symptoms (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Febuxostat 80 mg QD (N=267) | Febuxostat 120 mg QD (N=269) | Febuxostat 240 mg QD (N=134) | Allopurinol QD (N=268) | Placebo QD (N=134)
Diarrhoea (Excluding Infective) (Gastrointestinal disorders) | 16 | 19 | 18 | 17 | 11
Gastrointestinal & Abdominal Pains, Excluding Oral,Throat (Gastrointestinal disorders) | 5 | 7 | 8 | 6 | 3
Nausea and Vomiting Symptoms (Gastrointestinal disorders) | 11 | 10 | 8 | 6 | 5
Influenza Viral Infections (Infections and infestations) | 11 | 13 | 7 | 10 | 6
Upper Respiratory Tract Infections (Infections and infestations) | 39 | 52 | 27 | 52 | 21
Non-Site Specific Injuries NEC (Injury, poisoning and procedural complications) | 11 | 9 | 9 | 8 | 3
Liver Function Analyses (Investigations) | 17 | 10 | 6 | 15 | 3
Joint Related Signs and Symptoms (Musculoskeletal and connective tissue disorders) | 17 | 23 | 7 | 20 | 7
Muscle Related Signs and Symptoms NEC (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 1 | 7
Musculoskeletal and Connective Tissues Signs and Symptoms NEC (Musculoskeletal and connective tissue disorders) | 23 | 24 | 14 | 27 | 13
Headache NEC (Nervous system disorders) | 14 | 14 | 12 | 19 | 7
Neurological Signs and Symptoms NEC (Nervous system disorders) | 5 | 5 | 9 | 6 | 2
Vascular Hypertensive Disorders NEC (Vascular disorders) | 13 | 6 | 6 | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.